CLINICAL TRIAL: NCT02366897
Title: Extrapyramidal Side-Effects in Antipsychotic Drug Therapeutics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SensorPen.v.1.0
Record Dates: First submitted 2015-02-05; First posted 2015-02-19 (Estimated); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Drug-induced Extrapyramidal Side Effects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tolerability and sensitivity (Other): Stage 1: tolerability as per study design Stage 2: sensitivity as per study design - either quetiapine or risperidone. The intervention is the use of the Manus sensor pen
  Interventions: Device: Manus Sensor Pen

INTERVENTIONS:
Device: Manus Sensor Pen — Manus Sensor Pen as made by Manus Neurodynamica Ltd

SUMMARY:
The project is aimed at addressing the fundamental issue in antipsychotic therapeutics -the balance between mental state benefits and neurological risks.The latter cannot be overestimated and clinical skills in themselves are inadequately sensitive to refine practice. With all current and "pipeline" antipsychotics based on central dopamine blockade, there is little prospect that therapeutics can be improved by advances in pharmacology alone.

The project uses, for the first time, technology that is not only simple, real-life and user-friendly but "modern" and socially held in high regards. The proposal depends on patients receiving antipsychotic medication where clinically indicated. At all times, subjects will receive clinically-indicated therapy. The major ethical issue will relate to the issue of informed consent in those suffering from major psychiatric disorder. This is a routine consideration in psychiatric practice and the investigators will seek guidance on this from the Consultant Psychiatrist responsible for potential participants and would not proceed with initial approaches in cases of doubt or absence of capacity.

This is a pilot/feasibility study with no intention to utilise the data for commercialisation of the device or to expand the CE (Conformité Européenne) marking.

DETAILED DESCRIPTION:
The proposed methodology is based on use of a computer tablet and modified pen. While these instrumental elements are common-place and widely accepted in modern life, they are not so in the context of formal clinical assessment of motor function in psychiatric patients. They are also novel to clinicians. The first stage will involve recruitment of 20 patients i) under the age of 50 (to reduce the likelihood of idiopathic Parkinson's disease): ii) of mixed, balanced genders: iii) right-handed: iv) basic writing competence: v) English as first language: vi) suffering from an acute psychotic episode. These subjects will have been on stable doses of antipsychotic medication of any sort for at least 2 weeks. Patients will be seated in a comfortable writing position at a table and presented with a graphic tablet and a modified digitizer pen with a wired connection to an operator computer. The assessor will sit slightly behind and to one side out of the subject's view. To familiarise subjects with the technique, they will be asked to a) draw repetitive overlaid circles b) write their name and address, at a speed comfortable to them. They will then be asked to produce the 8 character 'el' text sequence ('elelelel') 10 times and to write a short, standard sentence : "Today is a nice day for the time of year". The examiner will then say to the subject the nursery rhyme, 'Mary had a little lamb...etc" and ask the subject to write it spontaneously from memory. Finally, they will be asked to copy a standard short paragraph from a written page. On conclusion, they will be asked to complete a brief 10cm line, Likert scale of satisfaction, assessing the test situation as 'easy/difficult: 'pleasurable/non-pleasurable':'acceptable/non-acceptable'.

PREDICTION : participants will find the procedures easy, pleasurable and acceptable

2 groups of 10 patients, complying with criteria i)-vi) above, but who have not been exposed to antipsychotic medication for at least 3 months (oral formulations) or 6 months (depot formulations) but in whom antipsychotic medication is now indicated. Groups will comprise consecutive consenting patients prescribed one of two commonly utilised antipsychotics : the high potency, risperidone, and the low potency, quetiapine. Dosages will be determined clinically by the responsible medical officers who will be asked to maintain a standard pattern of escalations : twice weekly and within the first 2 weeks of exposure (but not dose restricted). They will also be asked to avoid additional medications for drug-induced parkinsonism though these may be used on an as required 'rescue' basis. Other medications can be utilised as clinical need determines. Following informed consent, and prior to initiation of treatment, subjects will undertake baseline clinical assessments comprising : a standardised assessment of mental state (Positive and Negative Symptom Scale - PANSS); a standard clinical evaluation of extrapyramidal neurological status (the Extrapyramidal Symptom Rating Scale - ESRS); a standard questionnaire of subjective state (the Subjective Well-Being on Neuroleptics Scale - SWNS - designed to pick up later potential medication effects). They will then complete the instrumental component as above. Assessments will be completed twice weekly during the escalation phase (2 weeks) and weekly thereafter (up to 4 weeks) on the day before increases are implemented.

PREDICTION : instrumental methods will prove highly sensitive to the development of extrapyramidal side-effects and significantly more so than the standard clinical examination: AND : extrapyramidal effects will significantly precede the onset of antipsychotic efficacy

ELIGIBILITY:
Inclusion Criteria:

* Patients with an acute psychotic illness requiring admission to hospital
* Medications are deemed necessary for appropriate clinical management
* English as a first language
* Under the age of 50 years (to reduce the likelihood of idiopathic Parkinson's disease)
* Right-handed
* Mixed, balanced genders
* Basic writing competence
* No previous neurological disease

Exclusion Criteria:

* Lack of capacity as deemed by their Consultant Psychiatrist
* Under 18 years of age
* Over 50 years of age
* Recent use of psychostimulant drugs
* Previous neurological disease
* English not a first language
* Left handed
* Previous neurological condition
* For Stage 2: antipsychotic medication orally in the previous 3 months or by depot injection in the previous 6 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Acceptability to patients with acute psychotic illnesses using the Likert scale of satisfaction, assessing the test situation as 'easy/difficult: 'pleasurable/non-pleasurable':'acceptable/non-acceptable' | Stage 1 - One assessment for each patient, allow up to 4 weeks to recruit
Earlier onset (by >1 week) of parkinsonism assessed by micrographic changes compared to standard clinical examination as detected by the Manus sensor pen | Stage 2 - each patient shall be in the study for 6 weeks. Allow up to 6 months to recruit.

SECONDARY OUTCOMES:
Sensitivity: prevalence of parkinsonism at different criteria from rating scale parameters as detailed in "description" section below. | Stage 2 - each patient shall be in the study for 6 weeks. Allow up to 6 months to recruit.
  A standardised assessment of mental state (Positive and Negative Symptom Scale - PANSS); a standard clinical evaluation of extrapyramidal neurological status (the Extrapyramidal Symptom Rating Scale - ESRS); a standard questionnaire of subjective state (the Subjective Well-Being on Neuroleptics Scale - SWNS - designed to pick up later potential medication effects)

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom